CLINICAL TRIAL: NCT03526601
Title: Screening Of Adult urBan pOpulation To diAgnose Heart Failure
Acronym: SOBOTA-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital Murska Sobota (Other)
Collaborators: Roche Pharma AG (Industry); Slovenian Research Agency (Other); Murska Sobota Municipiality (Unknown); Community Health Center Murska Sobota (Unknown)
Responsible Party: Principal Investigator, Mitja Lainscak, Professor of Internal Medicine, General Hospital Murska Sobota
Other Study IDs: SBMS001
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
Keywords: heart failure; prevalence
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NT-proBNP, echocardiography — screening

SUMMARY:
Screening Of adult urBan pOpulation To diAgnose Heart Failure (SOBOTA-HF) is a cross-sectional prevalence study in a representative sample of Murska Sobota residents aged 55 years or more. Individuals will be invited to participate in a screening with NT-proBNP. All subjects with NT-proBNP ≥ 125 pg/mL will be invited for a diagnostic visit that will include history and physical examination, electrocardiogram, echocardiography, ankle brachial index, pulmonary function tests, body composition measurement, physical performance tests and questionnaires. To validate the screening procedure, a control group (NT-proBNP < 125 pg/mL) will undergo same diagnostic evaluation. An external center will validate echodardiography exams and the HF diagnosis will be adjudicated within an independent HF expert panel. Overall and age specific HF prevalence will be calculated in individuals ≥ 55 years and extrapolated to the whole population.

ELIGIBILITY:
Inclusion Criteria:

* age >55
* living in Murska Sobota
* part of representative sample as selected by Statistical Office of the Republic of Slovenia

Exclusion Criteria:

NONE.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60% of Murska Sobota residents aged 55 years or more
Sampling Method: Probability Sample
Enrollment: 2861 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
heart failure diagnosis as per 2016 ESC guidelines | at diagnostic visit

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainscak, MD, PhD, Principal Investigator — General Hospital Murska Sobota
Locations (1):
- General Hospital Murska Sobota, Murska Sobota, Slovenia

IPD SHARING:
Plan to Share IPD: No